CLINICAL TRIAL: NCT03891849
Title: Macro and Microcirculatory Effects of the Combination of Norepinephrine and Octreotide for the Treatment of Cirrhotic Patients With Hemorrhagic Shock
Acronym: HemodyNoOc
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participant enrolled. Equipment unvailable.
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0016
Record Dates: First submitted 2019-03-22; First posted 2019-03-27 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Haemorrhagic Shock; Variceal Hemorrhage
Keywords: microcirculation; octreotide; norepinephrine; Variceal Hemorrhage; Haemorrhagic Shock
MeSH Terms: conditions — Shock, Hemorrhagic | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- octreotide (25 µg/hour) perfusion (Experimental): octreotide (25 µg/hour) plus norepinephrine will be administered for patient with haemorrhagic shock after variceal bleeding during 2 to 5 days according recommendations and regular protocol in the medical unit
  Interventions: Drug: Octreotide Injection

INTERVENTIONS:
Drug: Octreotide Injection — Patients admitted in intensive care unit after variceal hemorrhage treated with norepinephrine perfusion will received an additional octreotide perfusion during one hour.

SUMMARY:
Octreotide is used to decrease portal pressure of cirrhotic patients admitted for variceal bleeding. When patients are in haemorrhagic shock, the recommended drug to increase arterial pressure is norepinephrine. Microcirculatory effects of octreotide when it is added to noradrenaline has not been investigated yet. The aim of the study is to evaluate the effect of octreotide plus norepinephrine for patient with haemorrhagic shock after variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years old
* patient with liver cirrhosis
* patient with haemorrhagic shock due to variceal bleeding
* patient with an arterial blood pressure less than 65 mmHg despite
* patient able to express consent
* signed written informed consent form
* patient covered by national health insurance

Exclusion Criteria:

* patient less than 18 years old
* patient non covered by national health insurance
* pregnant or breast feeding patent
* known octreotide allergy
* cardiac arrest because of shock
* refused consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of microcirculatory flow index | one hour after octreotide perfusion
  microcirculatory flow index will be measured with sidestream dark field handheld microscope. Baseline is before octreotide perfusion. Flow characteristics of the microvasculature will be quantified using the microcirculatory flow index (MFI) according to the recommendations from the consensus on microcirculatory imaging by De Backer et al. This index will be calculated after the image will be divided into four quadrants, and the predominant type of flow (absent = 0, intermittent = 1, sluggish = 2, abnormal = 3, and hyperdynamic = 4) would be estimated in the vessels smaller than 25 μm by the operator. The final MFI score is a value obtained from the average score of the four areas.
Change from baseline of microcirculatory flow index | 2 hours after octreotide perfusion
  microcirculatory flow index will be measured with sidestream dark field handheld microscope. Baseline is before octreotide perfusion. Flow characteristics of the microvasculature will be quantified using the microcirculatory flow index (MFI) according to the recommendations from the consensus on microcirculatory imaging by De Backer et al. This index will be calculated after the image will be divided into four quadrants, and the predominant type of flow (absent = 0, intermittent = 1, sluggish = 2, abnormal = 3, and hyperdynamic = 4) would be estimated in the vessels smaller than 25 μm by the operator. The final MFI score is a value obtained from the average score of the four areas.
Change from baseline of microcirculatory flow index | 6 hours after octreotide perfusion
  microcirculatory flow index will be measured with sidestream dark field handheld microscope. Baseline is before octreotide perfusion. Flow characteristics of the microvasculature will be quantified using the microcirculatory flow index (MFI) according to the recommendations from the consensus on microcirculatory imaging by De Backer et al. This index will be calculated after the image will be divided into four quadrants, and the predominant type of flow (absent = 0, intermittent = 1, sluggish = 2, abnormal = 3, and hyperdynamic = 4) would be estimated in the vessels smaller than 25 μm by the operator. The final MFI score is a value obtained from the average score of the four areas.
Change from baseline of microcirculatory flow index | 12 hours after octreotide perfusion
  microcirculatory flow index will be measured with sidestream dark field handheld microscope. Baseline is before octreotide perfusion. Flow characteristics of the microvasculature will be quantified using the microcirculatory flow index (MFI) according to the recommendations from the consensus on microcirculatory imaging by De Backer et al. This index will be calculated after the image will be divided into four quadrants, and the predominant type of flow (absent = 0, intermittent = 1, sluggish = 2, abnormal = 3, and hyperdynamic = 4) would be estimated in the vessels smaller than 25 μm by the operator. The final MFI score is a value obtained from the average score of the four areas.
Change from baseline of microcirculatory flow index | 24 hours after octreotide perfusion
  microcirculatory flow index will be measured with sidestream dark field handheld microscope. Baseline is before octreotide perfusion. Flow characteristics of the microvasculature will be quantified using the microcirculatory flow index (MFI) according to the recommendations from the consensus on microcirculatory imaging by De Backer et al. This index will be calculated after the image will be divided into four quadrants, and the predominant type of flow (absent = 0, intermittent = 1, sluggish = 2, abnormal = 3, and hyperdynamic = 4) would be estimated in the vessels smaller than 25 μm by the operator. The final MFI score is a value obtained from the average score of the four areas.

SECONDARY OUTCOMES:
percentage of perfused vessels | before and one hour after octreotide perfusion
  percentage of perfused vessels will be measured with sidestream dark field handheld microscope
percentage of perfused vessels | 2 hours after octreotide perfusion
  percentage of perfused vessels will be measured with sidestream dark field handheld microscope
percentage of perfused vessels | 6 hours after octreotide perfusion
  percentage of perfused vessels will be measured with sidestream dark field handheld microscope
percentage of perfused vessels | 12 hours after octreotide perfusion
  percentage of perfused vessels will be measured with sidestream dark field handheld microscope
percentage of perfused vessels | 24 hours after octreotide perfusion
  percentage of perfused vessels will be measured with sidestream dark field handheld microscope
functional capillary density | before and one hour after octreotide perfusion
  functional capillary density will be measured with sidestream dark field handheld microscope
functional capillary density | 2 hours after octreotide perfusion
  functional capillary density will be measured with sidestream dark field handheld microscope
functional capillary density | 6 hours after octreotide perfusion
  functional capillary density will be measured with sidestream dark field handheld microscope
functional capillary density | 12 hours after octreotide perfusion
  functional capillary density will be measured with sidestream dark field handheld microscope
functional capillary density | 24 hours after octreotide perfusion
  functional capillary density will be measured with sidestream dark field handheld microscope
Mean arterial pressure | before and one hour after octreotide perfusion
  Mean arterial pressure
Mean arterial pressure | 2 hours after octreotide perfusion
  Mean arterial pressure
Mean arterial pressure | 6 hours after octreotide perfusion
  Mean arterial pressure
Mean arterial pressure | 12 hours after octreotide perfusion
  Mean arterial pressure
Mean arterial pressure | 24 hours after octreotide perfusion
  Mean arterial pressure
heart rate | before and one hour after octreotide perfusion
  heart rate
heart rate | 2 hours after octreotide perfusion
  heart rate
heart rate | 6 hours after octreotide perfusion
  heart rate
heart rate | 12 hours after octreotide perfusion
  heart rate
heart rate | 24 hours after octreotide perfusion
  heart rate
ejection fraction | before and one hour after octreotide perfusion
  ejection fraction
ejection fraction | 2 hours after octreotide perfusion
  ejection fraction
ejection fraction | 6 hours after octreotide perfusion
  ejection fraction
ejection fraction | 12 hours after octreotide perfusion
  ejection fraction
ejection fraction | 24 hours after octreotide perfusion
  ejection fraction

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Malaquin, Dr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No